CLINICAL TRIAL: NCT00737165
Title: A Community Intervention Trial of Multimodal Suicide Prevention Program in Japan (NOCOMIT-J)
Acronym: NOCOMIT-J
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Japan Foundation for Neuroscience and Mental Health (Other)
Collaborators: National Center of Neurology and Psychiatry, Japan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: J-MISP-02; UMIN000000460 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Suicide
Keywords: Suicide, Prevention; Community
MeSH Terms: conditions — Suicide; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multimodal community intervention (Experimental): Multimodal suicide prevention program
  Interventions: Behavioral: Multimodal suicide prevention program
- Community intervention as usual (Active Comparator): Suicide prevention program as usual
  Interventions: Behavioral: Suicide prevention program as usual

INTERVENTIONS:
Behavioral: Multimodal suicide prevention program — A community intervention of multimodal suicide prevention program includes following components:
  1. Building support networks for suicide prevention and mental health promotion in public health system
  2. Primary prevention of suicide and suicide related behaviors
  3. Secondary prevention of suicide and suicide related behaviors
  4. Tertiary prevention; after care for suicide survivors
  5. Suicide prevention targeting for people with substance/alcohol- related disorders , schizophrenia and other mental health disorders
  6. Suicide prevention targeting for people with work-related problems
  Arms: Multimodal community intervention
Behavioral: Suicide prevention program as usual — Usual suicide prevention program
  Arms: Community intervention as usual

SUMMARY:
1. The primary goal for this study is to examine the effectiveness of community-based multimodal intervention program for suicide prevention in relatively high suicide rate region compared to control region.
2. The secondary goal for this study is to explore the effectiveness of community-based multimodal intervention program for suicide prevention in the highly populated regions. In addition, we examine the effectiveness of the prevention program in the all regions combined.

DETAILED DESCRIPTION:
Suicide is a major public health problem and the number of suicide victims has exceeded 30,000 a year since 1998 in Japan. Suicide rate is almost 25/100,000, which are remarkably high numbers among advanced countries. To examine the effectiveness of community-based multimodal intervention program for suicide prevention, a trial by J-MISP (Japanese Multimodal Intervention Trials for Suicide Prevention). This research project is one of the strategic research projects funded by The Japanese Ministry of Health, Labor and Welfare.

ELIGIBILITY:
Inclusion Criteria:

* Areas which meet the following criteria are eligible for this study;

  * An area with firm support from local government and other organizations to conduct this multimodal suicide prevention program
  * An area capable to select intervention and control regions
  * An area capable to follow the data collection procedure described in the protocol
  * An area with comparable baseline data on suicide attempts rate in intervention and control region
  * An area with comparable baseline data on demographics in intervention and control region

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1951060 (Actual)
Dates: Start 2006-07; Primary Completion 2009-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Incidence of suicide attempts (completed suicides and suicide attempts except mild case ) | 3.5years

SECONDARY OUTCOMES:
Incidence of completed suicides | 3.5years
Incidence of suicide attempts | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Ono, MD,PhD, Principal Investigator — Keio University
Locations (7):
- Japan (7):
  - Akita region group, Akita, Akita
  - Aomori region gruop, Aomori, Aomori
  - Chiba region group, Ichikawa, Chiba
  - Kita-Kyusyu region group, Kitakyushu, Fukuoka
  - Iwate region group, Morioka, Iwate
  - Minami Kyusyu region group, Kagoshima and Miyazaki, Kagoshima and Miyazaki
  - Sendai region group, Sendai, Miyagi

REFERENCES:
- [Background] Ono Y, Awata S, Iida H, Ishida Y, Ishizuka N, Iwasa H, Kamei Y, Motohashi Y, Nakagawa A, Nakamura J, Nishi N, Otsuka K, Oyama H, Sakai A, Sakai H, Suzuki Y, Tajima M, Tanaka E, Uda H, Yonemoto N, Yotsumoto T, Watanabe N. A community intervention trial of multimodal suicide prevention program in Japan: a novel multimodal community intervention program to prevent suicide and suicide attempt in Japan, NOCOMIT-J. BMC Public Health. 2008 Sep 15;8:315. doi: 10.1186/1471-2458-8-315. PMID 18793423
- [Background] Ono H, Awada S, Iida H, Ishida Y, Ishizuka N, Iwasa H, Kamei Y, Motohashi Y, Nakagawa A, Nakamura J, Nishi N, Otsuka K, Oyama H, Sakai A, Sakai H, Suzuki Y, Tajima M, Tanaka E, Uda E, Yonemoto N, Watanabe N. [Importance of area activities to prevent suicide and the involvement of NOCOMIT-J]. Seishin Shinkeigaku Zasshi. 2008;110(3):216-21. No abstract available. Japanese. PMID 18524043
- [Result] Ono Y, Sakai A, Otsuka K, Uda H, Oyama H, Ishizuka N, Awata S, Ishida Y, Iwasa H, Kamei Y, Motohashi Y, Nakamura J, Nishi N, Watanabe N, Yotsumoto T, Nakagawa A, Suzuki Y, Tajima M, Tanaka E, Sakai H, Yonemoto N. Effectiveness of a multimodal community intervention program to prevent suicide and suicide attempts: a quasi-experimental study. PLoS One. 2013 Oct 9;8(10):e74902. doi: 10.1371/journal.pone.0074902. eCollection 2013. PMID 24130673